CLINICAL TRIAL: NCT06279338
Title: A Clinical Study of Azacitidine Combined With BUCY2 Conditioning Regimen Before Allogeneic Hematopoietic Stem Cell Transplantation for Myelodysplastic Syndrome With Moderate High IPSS-M Score
Brief Title: A Novel Conditioning Regimen for Myelodysplastic Syndrome With Moderate High IPSS-M Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023] No.0969
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Molecular International Prognostic Scoring System (IPSS-M); Azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Azacitidine (Experimental): Combining azacitidine with classic BUCY2 regimen as conditioning regimen
  Interventions: Drug: Azacitidine Injection

INTERVENTIONS:
Drug: Azacitidine Injection — On the basis of the conventional transplantation treatment regimen, combining azacitidine injection with BUCY2 conditioning regimen (azacitidine 75 mg/m2/d for -11 days to -5 days, cytarabine 2 g/m2 q12h for -8 days to -7 days, cyclophosphamide 1.8 g/m2/d for -6 days to -5 days, busulfan 3.2 mg/kg/d for -4 days to -2 days)
  Other Names: Azacitidine

SUMMARY:
Figure out the Efficacy and Safety of Azacitidine Combined with BUCY2 Conditioning Regimen Before Allogeneic Hematopoietic Stem Cell Transplantation for Myelodysplastic Syndrome with Moderate High IPSS-M Score

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm clinical study, which plans to enroll 40 patients with high-risk myelodysplastic syndrome (MDS) to be given azacitidine (AZA) combined with busulfan and cyclophosphamide (BUCY2) conditioning regimen to evaluate 18-month progression-free survival (PFS), aiming to evaluate the efficacy and safety of azacitidine plus BUCY2 pretreatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand this study, voluntarily participate and sign the informed consent form
* Age equal or more than 18 years old
* Patients with moderate high-risk MDS with an IPSS-M score which is higher than 0
* Patients planning to undergo allogeneic hematopoietic stem cell transplantation, HCT-CI ≤ 3 or KPS ≥ 80%

Exclusion Criteria:

* Patients who refuse to participate in this clinical study
* Patients with central nervous system involvement
* Patients with HIV seropositive
* Patients with other serious medical conditions with a life expectancy of less than six months
* Patients with severe psychiatric or psychological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 18 months post-transplant, month | 18 months post-transplantation
  PFS is measured from the date of allo-HSCT to the date of relapse or death from any cause or the last follow-up for surviving patients.

SECONDARY OUTCOMES:
Overall survival (OS) at 18 months post-transplant, month | 18 months post-transplantation
  OS is defined as the time from allo-HSCT to the date of death from any cause or the last follow-up for surviving patients.

CONTACTS AND LOCATIONS:
Overall Officials: Linghui Xia, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology